CLINICAL TRIAL: NCT04950894
Title: Treating Obstructive Sleep Apnea Using Targeted Hypoglossal Neurostimulation
Acronym: OSPREY
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: LivaNova (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: LNS005
Record Dates: First submitted 2021-06-18; First posted 2021-07-06 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Obstructive Sleep Apnea; OSA; Apnea; Apnea, Obstructive; Apnea, Obstructive Sleep; Apnea+Hypopnea; Hypopnea, Sleep
Keywords: OSA; Snoring; Obstructive Sleep Apnea; CPAP; PAP
MeSH Terms: conditions — Sleep Apnea, Obstructive; Apnea; Sleep Apnea Syndromes; Snoring

STUDY DESIGN:
Intervention Model Description: All subjects are implanted and randomized. Stimulation treatment started at M1 for the Active group and M7 +1day for the Control group. Both groups followed through M13.
Who Masked: Investigator, Outcomes Assessor
Masking Description: PSG results are masked from the Investigator and Outcomes Assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Active (Active Comparator): HGN therapy activation at Month 1 - compared at Month 7 to Control group, continued stimulation through Month 13
  Interventions: Device: Hypoglossal Nerve Stimulation
- Control (Other): HGN therapy NOT activated at Month 1 - compared at Month 7 to Active group, stimulation will start at Month 7 + 1 Day and continue through Month 13
  Interventions: Device: Hypoglossal Nerve Stimulation

INTERVENTIONS:
Device: Hypoglossal Nerve Stimulation — Hypoglossal Nerve Stimulation started at Month 1 compared to no Stimulation (Control group will start stimulation at M7+1Day)

SUMMARY:
Multi-center, open-label, prospective, randomized clinical trial of the aura6000(R) System for the reduction of apnea and hypopneas in adult patients with moderate to severe obstructive sleep apnea who have failed or are unwilling to use positive airway pressure treatment.

DETAILED DESCRIPTION:
All qualifying subjects will be implanted. Subjects will be randomized 2:1 in favor of Stimulation therapy (Active Group). Randomization will occur following implant and prior to the Month 1 visit.

The Active group will start Stimulation therapy at Month 1. The Control group may continue with their current sleep apnea treatment until Month 7, and will receive Stimulation therapy beginning at Month 7 +1Day. (All subjects are excluded from use of PAP or surgical treatments after enrollment through Month 13)

Safety and efficacy will be evaluated at Month 7, and again at Month 13.

ELIGIBILITY:
Abbreviated: Additional criteria may apply:

Inclusion Criteria:

* Diagnosis of moderate to severe OSA
* Declines to use or does not tolerate PAP therapy

Exclusion Criteria:

* Respiratory, cardiac, renal disease or other co-morbid conditions
* BMI > 35 kg/m2
* Specific PSG criteria outlined in the protocol

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-07-27 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Rate of response to therapy when compared to no therapy for 6 months | Month 1 through Month 7
  The primary efficacy endpoint is to demonstrate that the AHI responder rate of subjects with the device stimulation activated (Active Group) is statistically significantly higher than the AHI responder rate of subjects with the device stimulation not activated (Control Group) at M7.
Rate of all serious adverse device/procedure related events from time of implant through month 7 | Month 1 through Month 7
  The primary safety endpoint is a descriptive evaluation of all reported serious adverse device/procedure related events (SADEs) through M7 for both groups. Relationship to procedure, device and study will be adjudicated by a Clinical Events Committee (CEC).

SECONDARY OUTCOMES:
Decrease in Oxygen Desaturation Index (Efficacy) | Baseline through Month 7
Change in Functional Outcomes of Sleep Questionnaire (Efficacy | Baseline through Month 7
Change in Epworth Sleepiness Scale (Efficacy) | Baseline through Month 7
Change in EQ-5D (Efficacy) | Baseline through Month 7
Change in PROMIS SDI/SRI (Efficacy) | Baseline through Month 7
Change in SF-36 (Efficacy) | Baseline through Month 7
Change in CGI-S/CGI-I (Efficacy) | Baseline through Month 7
Descriptive analysis of all reported Adverse Events (Safety) | Consent through Month 7

CONTACTS AND LOCATIONS:
Overall Officials: Atul Malhotra, MD, Principal Investigator — UCSD Pulmonary and Critical Care Medicine
Locations (20):
- United States (20):
  - University of Alabama At Birmingham, Birmingham, Alabama
  - Banner Health, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - Sacramento Ent, Roseville, California
  - Paul Schalch Lepe, Md/Silenso Clinic, San Diego, California
  - Sleep Medicine Specialists of South Florida, Miami, Florida
  - Morton Plant Mease Health Care, Safety Harbor, Florida
  - Advanced Ent Associates, Atlanta, Georgia
  - Norton Healthcare, Louisville, Kentucky
  - Alivation Research Llc, Lincoln, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Weill Cornell Medical College, New York, New York
  - Raleigh Neurology Associates, Pa, Raleigh, North Carolina
  - Penn State Health, Hershey, Pennsylvania
  - Philadelphia Ear, Nose and Throat Associates, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Bogan Sleep Consultants, Llc, Columbia, South Carolina
  - Houston Methodist, Houston, Texas
  - Epic Medical Research, Red Oak, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jacobowitz O, Schwartz AR, Lovett EG, Ranuzzi G, Malhotra A. Design and rationale for the treating Obstructive Sleep Apnea using Targeted Hypoglossal Nerve Stimulation (OSPREY) trial. Contemp Clin Trials. 2022 Aug;119:106804. doi: 10.1016/j.cct.2022.106804. Epub 2022 May 22. PMID 35613672